CLINICAL TRIAL: NCT05523271
Title: A Multi-center Control Study to Determine the Efficacy of CADEYE in Detecting Colon Polyps in Comparison to Standard of Care
Brief Title: A Multi Center Study Comparing the Efficacy of CAD EYE and the Standard of Care (White Light )
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Mostafa Ibrahim, Mostafa Ibrahim, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CADEYE
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer screening
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Diagnosis, Computer-Assisted

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing White Light Endoscopy (standard of care) (No Intervention): All subjects in Experimental Arm A will undergo SOC (white-light endoscopy).
- Patients undergoing CAD EYE endoscopy (Experimental): All subjects in Experimental Arm B will undergo CADEYE endoscopy.
  Interventions: Diagnostic Test: CAD EYE (Computer Aided Diagnosis ----?

INTERVENTIONS:
Diagnostic Test: CAD EYE (Computer Aided Diagnosis ----? — CADEYE is a CAD-e system (FUJIFILM) that enables real-time video processing at the same rate as the standard procedure and and allows a real time computer aided detection of polyps with high accuracy.
  Arms: Patients undergoing CAD EYE endoscopy

SUMMARY:
This study is to assess the sensitivity and added benefits of CADEYE compared to standard care (white-light) in detecting colon polyps in patients undergoing colonoscopy.

DETAILED DESCRIPTION:
Failure in polyp recognition is a major determinant for the high rate of missed colorectal neoplasms. In response, technological advances have paved the way for Computer-Aided Polyp Detection (CAD-e) systems. Artificial intelligence systems allow of real-time computer- aided detection of polyps with high-accuracy. CADEYE is a CAD-e system (FUJIFILM) that enables real-time video processing at the same rate as the standard procedure.

The data generated from this study will provide an estimate of the ADR throughout the Middle East as well as assess the accuracy of CADEYE in detecting adenomas in comparison to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years old subjects
* Subjects undergoing colonoscopy for the following: o Primary CRC screening

  * Post-polypectomy surveillance
  * Work up following FIT positivity
  * Symptoms/signs suspicions of CRC
* Subjects must be willing to give written informed consent for the trial

Exclusion Criteria:

* Unable to consent
* Contraindicated to undergo endoscopy
* Hospitalized patient
* Patients with the following conditions:

  * History of colon resection
  * History of CRC
  * Antithrombotic therapy precluding colon resection o Inflammatory Bowel Disease (IBD)
  * Familial Adenomatous Polyposis (FAP)
* Pregnant or lactating
* Poor bowel preparation: BBPS 0 or 1 in a segment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 1 year
  Adenoma detection rate is the primary end point which is the percentage of patients with at least 1 histologically proven adenoma or carcinoma.

SECONDARY OUTCOMES:
Adenomas detected per colonoscopy | 1 year
Proximal Adenoma detection rate | 1 year
Withdrawal time | 1 year
Non-neoplastic detection rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT05523271/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT05523271/ICF_001.pdf